CLINICAL TRIAL: NCT03212196
Title: Technical Strategies for Pancreatic Fistula Prevention After Pancreaticoduodenectomy in High-risk Pancreatic Remnant: a Risk-adjusted Randomized Controlled Trial
Brief Title: Technical Strategies for Pancreatic Fistula Prevention After Pancreaticoduodenectomy in High-risk Pancreatic Remnant
Acronym: PREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PREP 1041CESC
Record Dates: First submitted 2016-11-09; First posted 2017-07-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Fistula
Keywords: Pancreaticoduodenectomy; Pancreaticogastrostomy; Pancreaticojejunostomy; Stent; Transanastomotic drain
MeSH Terms: conditions — Pancreatic Fistula | interventions — Pancreaticojejunostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pancreaticogastrostomy (Active Comparator): Pancreaticogastrostomy with external drain
  Interventions: Procedure: Pancreaticogastrostomy with external drain
- Pancreaticojejunostomy (Active Comparator): Pancreaticojejunostomy with transanastomotic drain
  Interventions: Procedure: Pancreaticojejunostomy with transanastomotic drain

INTERVENTIONS:
Procedure: Pancreaticogastrostomy with external drain — Pancreatico-enteric anastomosis is provided according to the "Bassi technique", pancreatic remnant is pushed into the gastric cavity through a posterior gastrotomy. An externalized drain is placed into the main pancreatic duct.
  Arms: Pancreaticogastrostomy
Procedure: Pancreaticojejunostomy with transanastomotic drain — Pancreatico-enteric anastomosis is provided through a double-layer, duct-to-mucosa anastomosis with a transanastomotic externalized drain.
  Arms: Pancreaticojejunostomy

SUMMARY:
This trial will investigate what surgical technique between pancreaticogastrostomy and pancreaticojejunostomy with transanastomotic externalized drains is associated with the lowest rate of pancreatic fistula after pancreaticoduodenectomy in case of high-risk pancreatic remnants.

DETAILED DESCRIPTION:
Pancreatic fistula is the major determinant of outcome after pancreaticoduodenectomy. Several strategies to reduce the burden of this complication have been proposed in the last decade. A definite answer about what is the best technique to approach a high-risk pancreatic stump is still needed. Both pancreaticogastrostomy and pancreaticojejunostomy with transanastomotic externalized drains have been proposed in this setting, but often studies do not provide a reliable risk stratification and result are extremely variable.

The aim of this trial is to evaluate what surgical technique, between pancreaticogastrostomy and pancreaticojejunostomy with transanastomotic externalized drains, is associated with the lowest rate of pancreatic fistula in case of high-risk pancreatic remnants. Risk stratification will be provided through the Fistula Risk Score, a clinical risk score that has been extensively validated.

ELIGIBILITY:
Inclusion Criteria:

* All the patients undergoing pancreaticoduodenectomy (only Whipple or Traverso) for all kind of pancreatic disease (benign, malignant or premalignant).
* Patients able to give their informed consent

Exclusion criteria

* Informed consent withdrawal
* Impossibility to undergo surgery for any reason
* Use of glues or biological matrices to protect the anastomosis
* Fistula Risk Score < 7
* Post-operative octreotide analogues administration (only prophylactic use, therapeutic use allowed)
* Wrong randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Post-operative Pancreatic Fistula (POPF) | 30 days post-operative
  Presence of Amylase > 3 times the upper limit of normal in surgical drains at or by post-operative day 3 (POD) determining a clinically relevant change in patient's management

SECONDARY OUTCOMES:
POPF severity | 30 days post-operative
  POPF grade B and grade C rates
Length of Hospital Stay | 1 year
  calculated from the day of surgery to the day of discharge, adding up the days after a possible re-admission
Mortality | 90 days
  Death related to surgical morbidity
Post-Pancreatectomy Hemorrhage | 90 days
  As defined by the International Study Group for Pancreatic Surgery (ISGPS), grade A, B and C rates
Delayed Gastric Emptying | 90 days
  As defined by ISGPS, grade A, B and C rates
Biliary fistula | 90 days
  Output of bile from drains on or by POD 3, pancreaticojejunostomy leak should be ruled out
Gastrojejunal/Duodenojejunal fistula | 90 days
  Fistula from gastro/duodenojejunostomy
Abdominal abscess | 90 days
  Collection >5cm in size, containing gas bubbles, determining systemic signs of infection
Acute pancreatitis | 1 day post index surgery
  Altered serum amylase count on POD 0 or POD 1
Wound infection | 90 days
  Superficial and Deep Surgical Site Incisional Infection as defined by the Center for Disease Control and Prevention
Blood transfusions | 90 days
  Need and number of packed red blood cells transfused
Myocardial infarction | 90 days
  Myocardial necrosis
Acute Kidney Failure | 90 days
  Abrupt change in serum creatinine >1.5 baseline value
Pulmonary Embolism | 90 days
  Blood clots in the pulmonary arterial system
Pneumonia | 90 days
  Bacterial infection of the lungs
Respiratory insufficiency | 90 days
  Need for re-intubation
Urinary Tract Infection | 90 days
  Bacterial infection of the urinary tract
Cerebrovascular accidents | 90 days
  Stroke, hemorrhage, brain death
Reoperation | 90 days
  Need for new surgery due to severe morbidity
Readmission | 30 days after hospital discharge
  New admission within 30-days of discharge from hospital
Time-to-adjuvant therapy | 1 year
  Time form index operation to the beginning of adjuvant treatment (only for malignancy)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassi, MD, Principal Investigator — Università degli studi di Verona
Locations (1):
- Ospedale Policlinico GB Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers

REFERENCES:
- [Background] McMillan MT, Ecker BL, Behrman SW, Callery MP, Christein JD, Drebin JA, Fraker DL, Kent TS, Lee MK, Roses RE, Sprys MH, Vollmer CM Jr. Externalized Stents for Pancreatoduodenectomy Provide Value Only in High-Risk Scenarios. J Gastrointest Surg. 2016 Dec;20(12):2052-2062. doi: 10.1007/s11605-016-3289-6. Epub 2016 Oct 11. PMID 27730401
- [Background] Bassi C, Molinari E, Malleo G, Crippa S, Butturini G, Salvia R, Talamini G, Pederzoli P. Early versus late drain removal after standard pancreatic resections: results of a prospective randomized trial. Ann Surg. 2010 Aug;252(2):207-14. doi: 10.1097/SLA.0b013e3181e61e88. PMID 20622661
- [Background] Callery MP, Pratt WB, Kent TS, Chaikof EL, Vollmer CM Jr. A prospectively validated clinical risk score accurately predicts pancreatic fistula after pancreatoduodenectomy. J Am Coll Surg. 2013 Jan;216(1):1-14. doi: 10.1016/j.jamcollsurg.2012.09.002. Epub 2012 Nov 2. PMID 23122535
- [Background] Hallet J, Zih FS, Deobald RG, Scheer AS, Law CH, Coburn NG, Karanicolas PJ. The impact of pancreaticojejunostomy versus pancreaticogastrostomy reconstruction on pancreatic fistula after pancreaticoduodenectomy: meta-analysis of randomized controlled trials. HPB (Oxford). 2015 Feb;17(2):113-22. doi: 10.1111/hpb.12299. Epub 2014 Jul 7. PMID 25040921
- [Background] Wang SE, Chen SC, Shyr BU, Shyr YM. Comparison of Modified Blumgart pancreaticojejunostomy and pancreaticogastrostomy after pancreaticoduodenectomy. HPB (Oxford). 2016 Mar;18(3):229-35. doi: 10.1016/j.hpb.2015.09.007. Epub 2015 Nov 17. PMID 27017162
- [Derived] Andrianello S, Marchegiani G, Malleo G, Masini G, Balduzzi A, Paiella S, Esposito A, Landoni L, Casetti L, Tuveri M, Salvia R, Bassi C. Pancreaticojejunostomy With Externalized Stent vs Pancreaticogastrostomy With Externalized Stent for Patients With High-Risk Pancreatic Anastomosis: A Single-Center, Phase 3, Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):313-321. doi: 10.1001/jamasurg.2019.6035. PMID 32101272